CLINICAL TRIAL: NCT07012694
Title: A Prospective, Multicenter, Blinded, Randomized Controlled Trial Assessing the Diagnostic Yield and Tissue Adequacy of 22G Adapt Versus 22G Franseen Fine-Needle Biopsy for Solid Lesions Under Endoscopic Ultrasound Guidance
Brief Title: 22G-Adapt vs 22G-Franseen Needle Biopsy in EUS-Guided Tissue Acquisition of Solid Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First People's Hospital of Yunnan (Other); The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Bin Cheng, prof., Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Franseen FNB vs Adapt FNB 2025
Record Dates: First submitted 2025-05-25; First posted 2025-06-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Neoplasms; Mediastinal Neoplasms; Abdominal Neoplasm, Excluding Pancreas Neoplasm
Keywords: Endoscopic ultrasound; Fine-needle biopsy
MeSH Terms: conditions — Pancreatic Neoplasms; Mediastinal Neoplasms; Abdominal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 22G Franseen Needle Group (Experimental): 22G Franseen needles were adopted to acquire lesion tissues
  Interventions: Device: 22G Franseen Needle Group
- 22G Adapt Needle Group (Experimental): 22G Adapt needles were adopted to acquire lesion tissues
  Interventions: Device: 22G Adapt Needle Group

INTERVENTIONS:
Device: 22G Franseen Needle Group — Fine-needle-biopsy (22G Franseen, Boston Scientific, Winston-Salem, USA)
  Arms: 22G Franseen Needle Group
Device: 22G Adapt Needle Group — Fine-needle-biopsy (22G Adapt, Micro.Tech Endoscopy, Nanjing, China)
  Arms: 22G Adapt Needle Group

SUMMARY:
The investigators conduct a prospective, multicenter, blinded, randomized controlled trial to compare the diagnostic value and safety of the 22G Adapt needle versus the 22G Franseen needle for histopathological evaluation of solid lesions.

DETAILED DESCRIPTION:
Participants are randomized into two groups: the EUS-FNB-A group (22G Franseen needle) and the EUS-FNB-B group (22G Adapt needle). The primary endpoint is diagnostic accuracy for solid mass lesions. A non-inferiority design is adopted, with group A as the control. The significance level (α) is set at 0.025 (one-sided), with a type II error (β) of 0.15, providing a statistical power of 85%. Based on previous literature, the assumed diagnostic accuracy of the 22G Adapt FNB is 90%, compared to 92% for the 22G Franseen FNB, with a non-inferiority margin of -10%. Assuming a 1:1 allocation and accounting for a 20% dropout rate, 288 participants are planned for each group, totaling 576 participants.

Done by professional statistical people with randomized block grouping method and SAS 9.4 statistical software to generate randomized serial number（001-576）for the two groups in 1:1 manner. The serial numbers are the randomized grouping numbers for the trial patients, block capacity is 4, totally 144 randomized block. The randomized grouping will be generated in duplicate copies and sealed. One copy send to trial centers for patient allocating, and the another copy be saved by the trial applicant unit. Every trail centers will be responsible for the screening of qualified patients, rank them in visit time to get the randomized grouping number so as to determine them goes to the EUS-FNA or EUS-FNB.The research people and patients in all trial centers should not know the the randomized grouping number and relevant groups. The group name will be sealed under scratch card. Every trial patients will get a unique randomized number, and it will not change through out the whole trial.

Use the inclusion and exclusion criteria to observe the patients and do relative inspections, and confirm if the patients qualified or not to the trial. Record the result of last time test before the treatment. Although it is better to get the informed consent before doing all kinds of observation and tests, if for some reason, the medical imaging examination has completed, as long as the imaging examination was done within 3 weeks before the needle biopsy, it can still be collect as baseline data (imaging examination can be done at other hospitals, but the trial center should issue a new evaluation report 1 week before the patient join the trial group); other lab test items done at 2 weeks before the needle biopsy can still be collect as baseline data for pre-research use, but these tests should be done at the trail center hospital so as to guarantee the data trace ability.

The investigators will do the needle passes for 2 times for all of them:the 1 needle passes with Slow-Pull and the 2 needle passes with 5 mL wet suction. If no core tissues obtained or the operator/onsite pathologist determine insufficient specimen after the operations above, then remedy procedures will be done, the operator use proper puncture method to continue the remedy biopsy. After the first round of needle biopsy, if the trial patient cannot be diagnosed, by getting the agreement of the patient, the patient will be cross-over to another trial group and do needle biopsy again on the same lesion 1 week later with the method mentioned above. Without knowing the needle biopsy type, the cytologist and pathologist evaluate the specimen quality and make diagnosis. Every specimen will be independently evaluated and diagnosed by 2 experts. If the 2 experts have different judgments, then these two experts discuss together and make the final diagnose discussion. If the same sample has 2 or more cytology smear slides, than take the highest score slide as the result. Follow up (outpatient follow up or telephone follow up) the patients at 1 week, 12 weeks and 36 weeks after the needle biopsy and collect the patients clinical data and confirm their final diagnosis.

During the trial, if severe adverse event occurs, the trialed center must take immediate actions necessary to guarantee the trialed patients' safety. Once severe adverse event occurs, the researchers should inform the trial applicant and the trail center's ethics committee within 24 hours after the researchers gets to know the adverse event. And the researchers should also fax the report to State Food and Drug Administration of China and the local provincial food and drug administration. After receiving the report, the applicant should inform other clinical trial centers within 24 hours. All the severe adverse events should be filed at group leader medical center and other trial centers.

Case Report Form (CRF ) will be filled by the researchers, every involved patient must have the CRF filled. This will be audited by clinical monitor and handed over to data administrator to input and manage data, the first copy will be kept by the applicant, the second copy will go to the trial center, and the third copy will be kept by the trail researchers. The data input and management will be taken care by specially assigned person. In order to guarantee the data accuracy, data input will be done twice by two independent data administrators, by computerized and manual verifying, hand over the data to statistical experts to do blind check and statistic analyzing.For the questions and doubts within the case report form, the data administrator make Data Resolution Query (DRQ) and via the clinical monitor asking the researchers. The researchers will answer and feed back as soon as possible. According to the researchers answer, data administrator will do the data modifying, confirming or inputting, and when necessary send out DRQ again.After blind audition and confirming that the established data base is correct, major researchers, applicant and the statistic analyzing people lock the data. The locked data will not be changed, and the data base will be handed over to statistical analyzer to do the statistic analyze according to the statistic analyzing plan. Problems found after data locking can be modified during the statistic analyzing procedure.This will be done by specialized statistic analyzing people according to the predetermined statistic analyzing plan. The statistic analyze will be carried out according to intention principle confirmed full analysis set and per-protocol set principle. After completing the statistic analyzing, the statistic analyzer issue the statistic analysis report and send this to major researchers to write the study report.

Statistic analyzing plan:⑴ General principle:① all the statistic tests are use the two-tailed-test method, P<0.05 will be thought as the tested difference is statistical significance. ② the quantitative indicator description will calculate the Mean and Standard deviation. The classification indicator description will describe the cases and percentage of all types of cases. ⑵ Statistic analyzing method:① for the measurement data, compare it with the baseline value at selection period, use paired t-test or symbol rank sum test to compare with the before-after-difference within the group.② for the counting data, use x2 test or Fisher's exact test method to compare the groups. ⑶ Shedding analysis:Comparison of groups'total shedding rates and the shedding rates caused by adverse events will use x2 test or Fisher's exact test method. ⑷ The baseline value's equilibrium analysis: Use group t test or x2 test to compare the demography info and vital signs, disease history, and basic treatment and other indicators of baseline value, so as to measure the balance of the groups. The baseline evaluation will be done on Full Analysis Set (FAS) and Per-Protocol Set ( PPS). ⑸ Effectiveness analysis:The major indicator of effectiveness analysis is the diagnostic accuracy on malignant disease, and the indicators of second effectiveness include the percentage of Grade A specimen and complications rate etc. while the two groups rate and the Youden index comparison will use approximate normal Z test or use central effect x2 test.(6) Safety analysis:Use x2 test or Fisher's exact test to compare the adverse event/adverse reaction (include biopsy complications) rates between the groups. And use table to describe the adverse events during this trial project; the lab test results before and after the trial, the normal/abnormal changing condition and the relationship with this trial research when abnormal changes happened.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old and under 85 years old;
* Presence of a solid lesion greater than 1 cm in diameter, as identified by cross-sectional imaging (Magnetic Resonance Imaging, Computed Tomography or abdominal ultrasound), located in anatomical regions accessible via endoscopic ultrasound (EUS)-including but not limited to the pancreas, retroperitoneum, liver, mediastinum, or subepithelial layers of the gastrointestinal tract-where tissue acquisition is clinically indicated to establish a definitive histopathological diagnosis.;
* Must be able to receive examinations in the research center;
* Must be able to sign the informed consent.

Exclusion Criteria:

* Hemoglobin ≤8.0 g/dL;
* Pregnant women;
* Coagulation disorders(Platelet <50,000/mm3, International Normalized Ratio > 1.5);
* Took anticoagulants such as aspirin, warfarin in the latest week;
* Acute pancreatitis in the past two weeks;
* inability to safely perform Endoscopic Ultrasound-Guided Tissue Acquisition (eg, cardiorespiratory dysfunction, mental diseases, or drug addiction); refusal or inability to provide an informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
The histological diagnostic yields | up to 15 months
  The primary outcome measure of the study is to compare the histological diagnostic yield of EUS-guided fine-needle biopsy (EUS-FNB) using a 22G Franseen needle versus a 22G Adapt needle for both pancreatic and non-pancreatic solid lesions.

SECONDARY OUTCOMES:
The histological acquisition yields | up to 15 months
  Comparison of histological tissue acquisition adequacy between 22G Adapt and 22G Franseen needles in EUS-FNB of solid masses.
The cytological diagnosis yields | up to 15 months
  Comparison of cytological diagnostic yield between 22G Adapt and 22G Franseen needles in EUS-FNB of solid masses.
The Immunohistochemical (IHC) staining success rate | up to 15 months
  Comparison of successful IHC analysis rates of biopsy samples obtained using 22G Adapt versus 22G Franseen needles during EUS-FNB for solid masses.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cheng, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gkolfakis P, Crino SF, Tziatzios G, Ramai D, Papaefthymiou A, Papanikolaou IS, Triantafyllou K, Arvanitakis M, Lisotti A, Fusaroli P, Mangiavillano B, Carrara S, Repici A, Hassan C, Facciorusso A. Comparative diagnostic performance of end-cutting fine-needle biopsy needles for EUS tissue sampling of solid pancreatic masses: a network meta-analysis. Gastrointest Endosc. 2022 Jun;95(6):1067-1077.e15. doi: 10.1016/j.gie.2022.01.019. Epub 2022 Feb 4. PMID 35124072
- [Background] van Riet PA, Erler NS, Bruno MJ, Cahen DL. Comparison of fine-needle aspiration and fine-needle biopsy devices for endoscopic ultrasound-guided sampling of solid lesions: a systemic review and meta-analysis. Endoscopy. 2021 Apr;53(4):411-423. doi: 10.1055/a-1206-5552. Epub 2020 Aug 6. PMID 32583392
- [Background] Facciorusso A, Arvanitakis M, Crino SF, Fabbri C, Fornelli A, Leeds J, Archibugi L, Carrara S, Dhar J, Gkolfakis P, Haugk B, Iglesias Garcia J, Napoleon B, Papanikolaou IS, Seicean A, Stassen PMC, Vilmann P, Tham TC, Fuccio L. Endoscopic ultrasound-guided tissue sampling: European Society of Gastrointestinal Endoscopy (ESGE) Technical and Technology Review. Endoscopy. 2025 Apr;57(4):390-418. doi: 10.1055/a-2524-2596. Epub 2025 Feb 27. PMID 40015316
- [Background] Kovacevic B, Toxvaerd A, Klausen P, Larsen MH, Grutzmeier S, Detlefsen S, Karstensen JG, Brink L, Hassan H, Hogdall E, Vilmann P. Tissue amount and diagnostic yield of a novel franseen EUS-FNB and a standard EUS-FNA needle-A randomized controlled study in solid pancreatic lesions. Endosc Ultrasound. 2023 May-Jun;12(3):319-325. doi: 10.1097/eus.0000000000000007. Epub 2023 Jul 25. PMID 37693112
- [Background] Ashat M, Klair JS, Rooney SL, Vishal SJ, Jensen C, Sahar N, Murali AR, El-Abiad R, Gerke H. Randomized controlled trial comparing the Franseen needle with the Fork-tip needle for EUS-guided fine-needle biopsy. Gastrointest Endosc. 2021 Jan;93(1):140-150.e2. doi: 10.1016/j.gie.2020.05.057. Epub 2020 Jun 9. PMID 32526235
- [Background] Kurita A, Yasukawa S, Zen Y, Yoshimura K, Ogura T, Ozawa E, Okabe Y, Asada M, Nebiki H, Shigekawa M, Ikeura T, Eguchi T, Maruyama H, Ueki T, Itonaga M, Hashimoto S, Shiomi H, Minami R, Hoki N, Takenaka M, Itokawa Y, Uza N, Hashigo S, Yasuda H, Takada R, Kamada H, Kawamoto H, Kawakami H, Moriyama I, Fujita K, Matsumoto H, Hanada K, Takemura T, Yazumi S. Comparison of a 22-gauge Franseen-tip needle with a 20-gauge forward-bevel needle for the diagnosis of type 1 autoimmune pancreatitis: a prospective, randomized, controlled, multicenter study (COMPAS study). Gastrointest Endosc. 2020 Feb;91(2):373-381.e2. doi: 10.1016/j.gie.2019.10.012. Epub 2019 Oct 22. PMID 31654634
- [Background] Pouw RE, Barret M, Biermann K, Bisschops R, Czako L, Gecse KB, de Hertogh G, Hucl T, Iacucci M, Jansen M, Rutter M, Savarino E, Spaander MCW, Schmidt PT, Vieth M, Dinis-Ribeiro M, van Hooft JE. Endoscopic tissue sampling - Part 1: Upper gastrointestinal and hepatopancreatobiliary tracts. European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2021 Nov;53(11):1174-1188. doi: 10.1055/a-1611-5091. Epub 2021 Sep 17. PMID 34535035
- [Background] Cheng B, Zhang Y, Chen Q, Sun B, Deng Z, Shan H, Dou L, Wang J, Li Y, Yang X, Jiang T, Xu G, Wang G. Analysis of Fine-Needle Biopsy vs Fine-Needle Aspiration in Diagnosis of Pancreatic and Abdominal Masses: A Prospective, Multicenter, Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2018 Aug;16(8):1314-1321. doi: 10.1016/j.cgh.2017.07.010. Epub 2017 Jul 19. PMID 28733257
- [Background] Oh D, Kong J, Ko SW, Hong SM, So H, Hwang JS, Song TJ, Lee SK, Kim MH, Lee SS. A comparison between 25-gauge and 22-gauge Franseen needles for endoscopic ultrasound-guided sampling of pancreatic and peripancreatic masses: a randomized non-inferiority study. Endoscopy. 2021 Nov;53(11):1122-1129. doi: 10.1055/a-1369-8610. Epub 2021 Mar 2. PMID 33652495
- [Background] Gerke H, Rizk MK, Vanderheyden AD, Jensen CS. Randomized study comparing endoscopic ultrasound-guided Trucut biopsy and fine needle aspiration with high suction. Cytopathology. 2010 Feb;21(1):44-51. doi: 10.1111/j.1365-2303.2009.00656.x. Epub 2009 May 18. PMID 19456845
- [Background] Lee JK, Choi JH, Lee KH, Kim KM, Shin JU, Lee JK, Lee KT, Jang KT. A prospective, comparative trial to optimize sampling techniques in EUS-guided FNA of solid pancreatic masses. Gastrointest Endosc. 2013 May;77(5):745-51. doi: 10.1016/j.gie.2012.12.009. Epub 2013 Feb 21. PMID 23433878
- [Background] Crino SF, Conti Bellocchi MC, Di Mitri R, Inzani F, Rimbas M, Lisotti A, Manfredi G, Teoh AYB, Mangiavillano B, Sendino O, Bernardoni L, Manfrin E, Scimeca D, Unti E, Carlino A, Voiosu T, Mateescu RB, Fusaroli P, Lega S, Buscarini E, Pergola L, Chan SM, Lamonaca L, Gines A, Fernandez-Esparrach G, Facciorusso A, Larghi A. Wet-suction versus slow-pull technique for endoscopic ultrasound-guided fine-needle biopsy: a multicenter, randomized, crossover trial. Endoscopy. 2023 Mar;55(3):225-234. doi: 10.1055/a-1915-1812. Epub 2022 Aug 1. PMID 35915956